CLINICAL TRIAL: NCT06887218
Title: Randomized Phase II Trial of 5-Fluorouracil/Leucovorin (5FU/LV) in Combination With Regorafenib in Patients With Metastatic Colorectal Cancer
Brief Title: 5-Fluorouracil/Leucovorin (5FU/LV) in Combination With Regorafenib in Patients With Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Maen Abdelrahim, MD, PhD, Pharm.B, Section Chief Gastrointestinal Medical Oncology, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00038369 (HMCC-GI24-001)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Bevacizumab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5FU/LV in combination with regorafenib (Experimental): 5FU/LV will be administered to 38 patients as (LV [400 mg/m² IV over 120 minutes], followed by 5FU [400 mg/m² IV bolus then 2400 mg/m² IV infusion over 46 hours] in 2-week cycles) and regorafenib will be administered dose of 80-120 mg per day with weekly 40 mg per day increases to a maximum of 120 mg per day for 3 weeks on /1 week off until disease progression, up to 12 cycles of treatment.
  Interventions: Drug: Regorafenib (BAY 73-4506); Drug: 5FU/LV
- trifluridine-tipiracil (FTD-TPI) plus bevacizumab (Active Comparator): an additional 19 patients, will be given as FTD-TPI, administered orally, trice daily, at a starting dose of 35 mg/m2 of body-surface area, on days 1 through 5 and on days 8 through 12 every 28 days. Bevacizumab, at a dose of 5 mg per kilogram of body weight, will be administered intravenously on days 1 and 15. The 28-day treatment cycle continued until disease progression or unacceptable toxic effects occurred or consent was withdrawn, up to 12 cycles of treatment.
  Interventions: Drug: Bevacizumab; Drug: Trifluridine-tipiracil

INTERVENTIONS:
Drug: Regorafenib (BAY 73-4506) — Regorafenib will be administered a starting dose of 80 mg per day with weekly 40 mg per day increases to a maximum of 120 mg per day for 3 weeks on / 1 week off continued until disease progression or unacceptable toxic effects occurred or consent was withdrawn, up to 12 cycles of treatment.
  Arms: 5FU/LV in combination with regorafenib
Drug: 5FU/LV — 5FU/LV administered as (LV [400 mg/m² IV over 120 minutes], followed by 5FU [400 mg/m² IV bolus then 2400 mg/m² IV infusion over 46 hours] in 2-week cycles)
  Arms: 5FU/LV in combination with regorafenib
Drug: Bevacizumab — Bevacizumab, at a dose of 5 mg per kilogram of body weight, will be administered intravenously on days 1 and 15.
  Arms: trifluridine-tipiracil (FTD-TPI) plus bevacizumab
Drug: Trifluridine-tipiracil — FTD-TPI, administered orally, BID, at a starting dose of 35 mg/m2 of body-surface area, on days 1 through 5 and on days 8 through 12 every 28 days.
  Arms: trifluridine-tipiracil (FTD-TPI) plus bevacizumab

SUMMARY:
This is a non-inferiority randomized phase II trial investigating the efficacy and safety of 5FU/LV in combination with regorafenib for patients with metastatic colorectal cancer in the third-line setting.

Patients will be randomly assigned in a 2:1 ratio between 5FU/LV combined with regorafenib or trifluridine-tipiracil (FTD-TPI) plus bevacizumab.

Arm 1 (Treatment Arm) will consist of the 5FU/LV administered to 38 patients as (LV [400 mg/m² IV over 120 minutes], followed by 5FU [400 mg/m² IV bolus then 2400 mg/m² IV infusion over 46 hours] in 2-week cycles) and regorafenib will be administered dose of 80-120 mg per day with weekly 40 mg per day increases to a maximum of 120 mg per day for 3 weeks on /1 week off until disease progression, up to 12 cycles of treatment.

Arm 2 (Control Arm) received by an additional 19 patients, will be given as FTD-TPI, administered orally, BID, at a starting dose of 35 mg/m2 of body-surface area, on days 1 through 5 and on days 8 through 12 every 28 days. Bevacizumab, at a dose of 5 mg per kilogram of body weight, will be administered intravenously on days 1 and 15. The 28-day treatment cycle continued until disease progression or unacceptable toxic effects occurred or consent was withdrawn, up to 12 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Histopathological or cytologically confirmed metastatic CRC.
3. Failed second-line therapy for metastatic disease.
4. A minimum of one measurable disease per RECISTv1.1.
5. ECOG performance status of 0-2.
6. Life expectancy ≥6 months per treating physician or principal investigator.
7. Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
8. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

   a. Total bilirubin ≤ 10 x the upper limits of normal (ULN) b. Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer) c. Alkaline phosphatase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer) d. Serum creatinine ≤ 1.5 x the ULN e. International normalized ratio (INR)/ Partial thromboplastin time (PTT) ≤ 1.5 x ULN. (Subjects who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care.

   f. Platelet count ≥100000 /mm3, hemoglobin (Hb) ≥9 g/dL, absolute neutrophil count (ANC) ≥1500/mm3. Blood transfusion to meet the inclusion criteria will not be allowed.
9. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test. The definition of adequate contraception will be based on the judgment of the investigator.
10. Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 2 months after the last dose of study drug as outlined in Appendices 12.2
11. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
12. Subject must be able to swallow and retain oral medication.

Exclusion Criteria:

* 1. Hematology laboratory values of:

  1. Absolute neutrophil count ≤1000 cells/mm3
  2. Platelets ≤70,000 cells/mm3
  3. Hemoglobin ≤9 g/dL
  4. White blood count ≤3000 cells/mm3. 2. Hepatic laboratory values of aspartate transaminase or alanine aminotransferase:

  <!-- -->

  1. >5 × upper limits of normal (ULN) if the documented history of hepatic metastases; or
  2. >2.5 × ULN if no liver metastases are present. 3. Serum albumin <5.8 g/dL. 4. Total bilirubin >10 mg/dL. 5. Prothrombin time (PT) or international normalized ratio (INR) >1.5 × ULN. Note: Patients receiving therapeutic doses of anticoagulant therapy may be considered eligible if PT and INR are within the acceptable institutional therapeutic limits.

     6. Serum creatinine or serum urea >1.5 × ULN. 7. Estimated glomerular filtration rate <50 mL/min. 8. Positive pregnancy test, pregnant, or breastfeeding (female patients only). 9. Any other clinically significant laboratory abnormality that would compromise patient safety or the outcome of the study.

     10. Any clinically significant and/or uncontrolled cardiac-related abnormality that would compromise patient safety or the outcome of the study including, but not limited to:

  <!-- -->

  1. Arrhythmia
  2. Bradycardia
  3. Tachycardia
  4. Symptomatic valvular disease
  5. Symptomatic congestive heart failure is classified by New York Heart Association as Class III or IV
  6. Unstable angina pectoris. 11. Myocardial infarction within the past 6 months from the consent date. 12. Active bleeding diathesis. 13. Current complaints of persistent constipation or history of chronic constipation, bowel obstruction, or fecaloma within the past 6 months from the consent date.

     14. Known history and/or uncontrolled hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV)-1 or HIV-2 from the consent date.

     15. Active or recent (within 3 years) non-colorectal cancer malignancies, except for low-risk, cured cancers (e.g., squamous or basal cell carcinomas, in situ carcinomas, or others deemed non-significant by the investigator).

     16. Receipt of live, attenuated vaccine (e.g., intranasal influenza, measles, mumps, rubella, varicella) or close contact with someone who has received a live, attenuated vaccine within the past 1 month. Note: Influenza vaccine will be allowed if administered >21 days.

     17. Receipt of any investigation agent or study treatment within the past 30 days.

     18. Ongoing infection > Grade 2 NCI-CTCAE V5.0. 19. Symptomatic metastatic brain or meningeal tumors. 20. The presence of a non-healing wound, non-healing ulcer, or bone fracture. 21. Major surgical procedure or significant traumatic injury within 28 days before start of study medication 22. Renal failure that requires hemo-or peritoneal dialysis.

  <!-- -->

  1. Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study.

     23. Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE V5.0] on repeated measurement) despite optimal medical management.

     24. Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.

     25. Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment within 6 months of informed consent.

     26. Patients with any previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated ductal carcinoma in situ of the breast, curatively treated nonmelanoma skin carcinoma, noninvasive aerodigestive neoplasms, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before registration are allowed. All cancer treatments must be completed at least 3 years prior to registration.

     27. Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE V5.0 Grade 2 dyspnea).

     28. Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.

     29. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.

     30. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 57 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 5FU/LV in combination with regorafenib in metastatic colorectal cancer | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 18 months.
  Overall survival rate of patients with metastatic colorectal cancer treated with 5FU/LV in combination with regorafenib at 12 months.

SECONDARY OUTCOMES:
Progression-free survival rate of patients with metastatic colorectal cancer treated with 5FU/LV in combination with regorafenib | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 18 months.
  Progression-free survival rate of patients with metastatic colorectal cancer treated with 5FU/LV in combination with regorafenib according to RECIST v1.1 criteria.
Duration of the response of 5FU/LV in combination with regorafenib in third-line metastatic colorectal cancer patients | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 18 months.
  Duration of the response of 5FU/LV in combination with regorafenib in third-line metastatic colorectal cancer patients from onset of response to progression or death, whichever occurs earlier according to RECIST v1.1 criteria and investigator's tumor assessment.
Safety and tolerability of 5FU/LV in combination with regorafenib. | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study, whichever came first, assessed up to 13 months.
  To determine the safety and tolerability of 5FU/LV in combination with regorafenib (determined by diseases progression, unacceptable toxicity, and physician's discretion).

OTHER OUTCOMES:
Changes in health-related quality of life | From baseline to months 6 and 12
  Changes in health-related quality of life from baseline to months 6 and 12, as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 scores range from 0 to 100. For global health status/quality of life and functional scales (e.g., physical, role, emotional, cognitive, social), higher scores indicate better outcomes (improved quality of life or functioning). For symptom scales/items (e.g., fatigue, pain, nausea/vomiting), higher scores indicate worse outcomes (more severe symptoms).
Time to treatment failure of 5FU/LV in combination with regorafenib | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study, whichever came first, assessed up to 18 months.
  Time to treatment failure of 5FU/LV in combination with regorafenib (determined by diseases progression, unacceptable toxicity, and physician's discretion).

CONTACTS AND LOCATIONS:
Overall Officials: Maen Abdelrahim, MD, PhD, Pharm D, Principal Investigator — The Methodist Hospital Research Institute; Abdullah Esmail, MD, Study Director — Houston Methodist Neal Cancer Center
Locations (1):
- Houston Methodist Neal Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marks EI, Tan C, Zhang J, Zhou L, Yang Z, Scicchitano A, El-Deiry WS. Regorafenib with a fluoropyrimidine for metastatic colorectal cancer after progression on multiple 5-FU-containing combination therapies and regorafenib monotherapy. Cancer Biol Ther. 2015;16(12):1710-9. doi: 10.1080/15384047.2015.1113355. PMID 26561209
- [Background] Diez M, Teule A, Salazar R. Gastroenteropancreatic neuroendocrine tumors: diagnosis and treatment. Ann Gastroenterol. 2013;26(1):29-36. PMID 24714698
- [Background] Haque E, Muhsen IN, Esmail A, Umoru G, Mylavarapu C, Ajewole VB, Abdelrahim M. Case report: Efficacy and safety of regorafenib plus fluorouracil combination therapy in the treatment of refractory metastatic colorectal cancer. Front Oncol. 2022 Dec 15;12:992455. doi: 10.3389/fonc.2022.992455. eCollection 2022. PMID 36620581
- [Background] Pfeiffer P, Yilmaz M, Moller S, Zitnjak D, Krogh M, Petersen LN, Poulsen LO, Winther SB, Thomsen KG, Qvortrup C. TAS-102 with or without bevacizumab in patients with chemorefractory metastatic colorectal cancer: an investigator-initiated, open-label, randomised, phase 2 trial. Lancet Oncol. 2020 Mar;21(3):412-420. doi: 10.1016/S1470-2045(19)30827-7. Epub 2020 Jan 27. PMID 31999946
- [Background] Kuboki Y, Nishina T, Shinozaki E, Yamazaki K, Shitara K, Okamoto W, Kajiwara T, Matsumoto T, Tsushima T, Mochizuki N, Nomura S, Doi T, Sato A, Ohtsu A, Yoshino T. TAS-102 plus bevacizumab for patients with metastatic colorectal cancer refractory to standard therapies (C-TASK FORCE): an investigator-initiated, open-label, single-arm, multicentre, phase 1/2 study. Lancet Oncol. 2017 Sep;18(9):1172-1181. doi: 10.1016/S1470-2045(17)30425-4. Epub 2017 Jul 28. PMID 28760399
- [Background] Mayer RJ, Van Cutsem E, Falcone A, Yoshino T, Garcia-Carbonero R, Mizunuma N, Yamazaki K, Shimada Y, Tabernero J, Komatsu Y, Sobrero A, Boucher E, Peeters M, Tran B, Lenz HJ, Zaniboni A, Hochster H, Cleary JM, Prenen H, Benedetti F, Mizuguchi H, Makris L, Ito M, Ohtsu A; RECOURSE Study Group. Randomized trial of TAS-102 for refractory metastatic colorectal cancer. N Engl J Med. 2015 May 14;372(20):1909-19. doi: 10.1056/NEJMoa1414325. PMID 25970050
- [Background] Ishiguro M, Kotake K, Nishimura G, Tomita N, Ichikawa W, Takahashi K, Watanabe T, Furuhata T, Kondo K, Mori M, Kakeji Y, Kanazawa A, Kobayashi M, Okajima M, Hyodo I, Miyakoda K, Sugihara K. Study protocol of the B-CAST study: a multicenter, prospective cohort study investigating the tumor biomarkers in adjuvant chemotherapy for stage III colon cancer. BMC Cancer. 2013 Mar 25;13:149. doi: 10.1186/1471-2407-13-149. PMID 23530572
- [Background] Nordic Gastrointestinal Tumor Adjuvant Therapy Group. Expectancy or primary chemotherapy in patients with advanced asymptomatic colorectal cancer: a randomized trial. J Clin Oncol. 1992 Jun;10(6):904-11. doi: 10.1200/JCO.1992.10.6.904. PMID 1588370
- [Background] Mohelnikova-Duchonova B, Melichar B, Soucek P. FOLFOX/FOLFIRI pharmacogenetics: the call for a personalized approach in colorectal cancer therapy. World J Gastroenterol. 2014 Aug 14;20(30):10316-30. doi: 10.3748/wjg.v20.i30.10316. PMID 25132748
- [Background] Bekaii-Saab TS, Ou FS, Ahn DH, Boland PM, Ciombor KK, Heying EN, Dockter TJ, Jacobs NL, Pasche BC, Cleary JM, Meyers JP, Desnoyers RJ, McCune JS, Pedersen K, Barzi A, Chiorean EG, Sloan J, Lacouture ME, Lenz HJ, Grothey A. Regorafenib dose-optimisation in patients with refractory metastatic colorectal cancer (ReDOS): a randomised, multicentre, open-label, phase 2 study. Lancet Oncol. 2019 Aug;20(8):1070-1082. doi: 10.1016/S1470-2045(19)30272-4. Epub 2019 Jun 28. PMID 31262657
- [Background] Demetri GD, Reichardt P, Kang YK, Blay JY, Rutkowski P, Gelderblom H, Hohenberger P, Leahy M, von Mehren M, Joensuu H, Badalamenti G, Blackstein M, Le Cesne A, Schoffski P, Maki RG, Bauer S, Nguyen BB, Xu J, Nishida T, Chung J, Kappeler C, Kuss I, Laurent D, Casali PG; GRID study investigators. Efficacy and safety of regorafenib for advanced gastrointestinal stromal tumours after failure of imatinib and sunitinib (GRID): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):295-302. doi: 10.1016/S0140-6736(12)61857-1. Epub 2012 Nov 22. PMID 23177515
- [Background] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Background] Apperley JF, Gardembas M, Melo JV, Russell-Jones R, Bain BJ, Baxter EJ, Chase A, Chessells JM, Colombat M, Dearden CE, Dimitrijevic S, Mahon FX, Marin D, Nikolova Z, Olavarria E, Silberman S, Schultheis B, Cross NC, Goldman JM. Response to imatinib mesylate in patients with chronic myeloproliferative diseases with rearrangements of the platelet-derived growth factor receptor beta. N Engl J Med. 2002 Aug 15;347(7):481-7. doi: 10.1056/NEJMoa020150. PMID 12181402
- [Background] Bergers G, Song S, Meyer-Morse N, Bergsland E, Hanahan D. Benefits of targeting both pericytes and endothelial cells in the tumor vasculature with kinase inhibitors. J Clin Invest. 2003 May;111(9):1287-95. doi: 10.1172/JCI17929. PMID 12727920
- [Background] Ferrara N. VEGF and the quest for tumour angiogenesis factors. Nat Rev Cancer. 2002 Oct;2(10):795-803. doi: 10.1038/nrc909. PMID 12360282
- [Background] Wilhelm SM, Dumas J, Adnane L, Lynch M, Carter CA, Schutz G, Thierauch KH, Zopf D. Regorafenib (BAY 73-4506): a new oral multikinase inhibitor of angiogenic, stromal and oncogenic receptor tyrosine kinases with potent preclinical antitumor activity. Int J Cancer. 2011 Jul 1;129(1):245-55. doi: 10.1002/ijc.25864. Epub 2011 Apr 22. PMID 21170960
- [Background] Prager GW, Taieb J, Fakih M, Ciardiello F, Van Cutsem E, Elez E, Cruz FM, Wyrwicz L, Stroyakovskiy D, Papai Z, Poureau PG, Liposits G, Cremolini C, Bondarenko I, Modest DP, Benhadji KA, Amellal N, Leger C, Vidot L, Tabernero J; SUNLIGHT Investigators. Trifluridine-Tipiracil and Bevacizumab in Refractory Metastatic Colorectal Cancer. N Engl J Med. 2023 May 4;388(18):1657-1667. doi: 10.1056/NEJMoa2214963. PMID 37133585
- [Background] Reddy TP, Khan U, Burns EA, Abdelrahim M. Chemotherapy rechallenge in metastatic colon cancer: A case report and literature review. World J Clin Oncol. 2020 Nov 24;11(11):959-967. doi: 10.5306/wjco.v11.i11.959. PMID 33312889